CLINICAL TRIAL: NCT02620098
Title: Effectiveness of a Handwriting Intervention With At-Risk Kindergarteners
Brief Title: Effectiveness of a Handwriting Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Principal Investigator, Beth Pfeiffer, Associate Professor, Temple University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hand01
Record Dates: First submitted 2015-11-18; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Developmental Dysgraphia
MeSH Terms: conditions — Agraphia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Size Matters Handwriting Program (Experimental): All participants were receiving educational support in the form of IEP and/or RtI tier 2 interventions, and were participating in a support classroom where those services where being delivered. The intervention group consisted of 23 kindergarten students comprising all students in two kindergarten support classrooms, one in each of two neighboring schools. All students in the group received the Size Matters Handwriting Program.
  Interventions: Other: Size Matters Handwriting Program
- Control (No Intervention): All participants were receiving educational support in the form of IEP and/or RtI tier 2 interventions, and were participating in a support classroom where those services where being delivered. The control group consisted of 12 kindergarteners comprising all students in a kindergarten support classroom at a third school. They received no additional interventions.

INTERVENTIONS:
Other: Size Matters Handwriting Program — The Size Matters Handwriting Program (Moskowitz, 2009) (SMHP) program incorporates principles grounded in motor learning theory, cognitive theory, and motivation theory. Children learn the importance of letter size by learning size 1 (capital and tall letters), size 2 (small letters) and size 3 letters (those that dive below the baseline) at different stages (Moskowitz, 2009). The intervention group received a total of 30 sessions of the SMHP, completed twice weekly over a 16 week period. Sessions lasted 30 minutes, and were led by an occupational therapist with training in the Size Matters Handwriting Program. All interventions were provided within the existing support classrooms. Each child had their own SMHP workbook.
  Arms: Size Matters Handwriting Program

SUMMARY:
The purpose of the study was to examine the effectiveness of an occupational therapy led handwriting intervention for special education and at-risk kindergarten students.

DETAILED DESCRIPTION:
In spite of the increased use of computers and tablets by children of younger and younger ages, handwriting remains an important skill for school success and continues to be a critical skill for elementary school students to acquire. Beginning writers still do most of their composing by hand, and difficulties with handwriting can have far-reaching effects on a child's self esteem and academic success.

This study examined the effectiveness of an occupational therapy led handwriting intervention for special education and at-risk kindergarten students. There is a tremendous need for studies examining the outcomes of handwriting instruction provided to the at-risk population, in order to determine whether outcomes are similar to those seen in the typically developing population. There is also a need for studies that examine outcomes in "real world" settings, in addition to those settings manipulated for experimental research. Such studies may not be as "clean" as those in classic experimental research, however it is imperative to examine outcomes in the settings that are occurring in today's schools. At-risk children are increasingly being provided intensive interventions under an RtI model, and children receiving special education services are increasingly being integrated into less restrictive settings, thus creating classroom environments with a wide variety of students needs.

The purpose of this study was to examine the outcomes of a handwriting intervention, the Size Matters Handwriting Program (SMHP), provided to kindergarten children currently receiving IEP or RtI interventions. This study attempted to answer the following research questions:

1. Will at-risk kindergarteners (those children receiving IEP or RtI support) participating in a 16 week, occupational therapy led handwriting SMHP intervention group demonstrate significantly greater improvements in handwriting legibility than children who do not receive the intervention?
2. Will at-risk kindergarteners, participating in a SMHP handwriting intervention, make significantly greater gains in the pre-reading skills of letter-name recognition and letter-sound recall, than students who do not receive the intervention?

The study incorporated a two group pre and post-test design. Both groups consisted of kindergarten students receiving IEP and/or RtI support. An occupational therapist provided biweekly group handwriting instruction using the Size Matters Handwriting Program to students in the intervention group (n = 23), while the control group (n=12) received the standard handwriting instruction.

ELIGIBILITY:
* Inclusion Criteria:

  * Kindergartners receiving educational support in the form of IEP and/or RtI tier 2 interventions
  * Must be in a support classroom where services are delivered
* Exclusion Criteria:

  * Children not in kindergarten
  * Children not receiving IEP or Rtl tier 2 interventions

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in the Test of Handwriting Skills-Revised (THS-R) after 16 weeks | Before and after 30 sessions completed twice a week for 16 weeks
  A standardized assessment of handwriting which can be administered to students ages six to 18 (Milone, 2007). There are ten subtests which include writing letters and numbers from memory, writing letters, numbers and words from dictation, copying letters, copying words, copying short sentences, and writing short words from dictation (Milone, 2007).

SECONDARY OUTCOMES:
Change in the North Dakota Title I Kindergarten Reading Standards Assessment (Letter Identification Subtest after 16 weeks | Before and after 30 sessions completed twice a week for 16 weeks
  The North Dakota Kindergarten Reading Standards Assessment is aligned with North Dakota State Standards and consists of a number of subtests including: letter identification, word recognition, concepts about print, and sentence dictation. The assessment was designed as a tool for teachers and educational in selecting Title I students or assessing student achievement.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Pfeiffer, PhD, Principal Investigator — Temple University

REFERENCES:
- [Background] Bradley R, Danielson L, Doolittle J. Response to intervention. J Learn Disabil. 2005 Nov-Dec;38(6):485-6. doi: 10.1177/00222194050380060201. PMID 16392688
- [Background] Case-Smith J, Holland T, Bishop B. Effectiveness of an integrated handwriting program for first-grade students: a pilot study. Am J Occup Ther. 2011 Nov-Dec;65(6):670-8. doi: 10.5014/ajot.2011.000984. PMID 22214111
- [Background] Case-Smith J, Holland T, Lane A, White S. Effect of a coteaching handwriting program for first graders: one-group pretest-posttest design. Am J Occup Ther. 2012 Jul-Aug;66(4):396-405. doi: 10.5014/ajot.2012.004333. PMID 22742687
- [Background] Case-Smith J, Weaver L, Holland T. Effects of a classroom-embedded occupational therapist-teacher handwriting program for first-grade students. Am J Occup Ther. 2014 Nov-Dec;68(6):690-8. doi: 10.5014/ajot.2014.011585. PMID 25397764
- [Background] Dunsmuir S, Blatchford P. Predictors of writing competence in 4- to 7-year-old children. Br J Educ Psychol. 2004 Sep;74(Pt 3):461-83. doi: 10.1348/0007099041552323. PMID 15296550
- [Background] Feder KP, Majnemer A. Handwriting development, competency, and intervention. Dev Med Child Neurol. 2007 Apr;49(4):312-7. doi: 10.1111/j.1469-8749.2007.00312.x. PMID 17376144
- [Background] Howe TH, Roston KL, Sheu CF, Hinojosa J. Assessing handwriting intervention effectiveness in elementary school students: a two-group controlled study. Am J Occup Ther. 2013 Jan-Feb;67(1):19-26. doi: 10.5014/ajot.2013.005470. PMID 23245779
- [Background] James KH, Engelhardt L. The effects of handwriting experience on functional brain development in pre-literate children. Trends Neurosci Educ. 2012 Dec;1(1):32-42. doi: 10.1016/j.tine.2012.08.001. PMID 25541600
- [Background] Ohl AM, Graze H, Weber K, Kenny S, Salvatore C, Wagreich S. Effectiveness of a 10-week tier-1 response to intervention program in improving fine motor and visual-motor skills in general education kindergarten students. Am J Occup Ther. 2013 Sep-Oct;67(5):507-14. doi: 10.5014/ajot.2013.008110. PMID 23968788
- [Background] Pfeiffer B, Rai G, Murray T, Brusilovskiy E. Effectiveness of the Size Matters Handwriting Program. OTJR (Thorofare N J). 2015 Apr;35(2):110-9. doi: 10.1177/1539449215573004. PMID 26460474